CLINICAL TRIAL: NCT02169349
Title: Advancing Monitoring of NSCLC Treated With Epidermal Growth Factor Receptor (EGFR)-Tyrosine Kinase Inhibitor (TKI) - Molecular Diagnosis on Circulating Tumor DNA
Brief Title: Molecular Diagnosis on Circulating Tumor DNA of Non-Small Cell Lung Cancer
Acronym: ANTiCIPe
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: 2014-A00426-41
Record Dates: First submitted 2014-06-04; First posted 2014-06-23 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2015-10

CONDITIONS: Stage IIIb and IV Non Small Cell Lung Cancer
MeSH Terms: interventions — High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Other: laboratory biomarker analysis
Other: Next Generation Sequencing
Genetic: DNA Analysis

SUMMARY:
The purpose of this study is to develop an ultra sensitive assay of mutation detection on circulating tumor DNA (ctDNA) for treatment, diagnosis and monitoring disease progression of Non-Small Cell Lung Cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Male or female aged >= 18 years
* Stage IIIb and IV Non Small Cell Lung Cancer histologically confirmed

Exclusion Criteria:

* Tissue and plasma samples can not be provided for mutation analysis
* Unwilling or unable to provide informed consent
* Any serious medical condition that would interfere with the subject's safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from patients receiving treatment for NSCLC at the Rennes Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-06; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Mutation profiling of circulating tumor DNA from plasma samples. | 1 year
  To evaluate the sensitivity of NGS to detect the genetic alterations in plasma tumor DNA.

SECONDARY OUTCOMES:
Quantity of circulating tumor DNA in serially collected plasma specimens. | 1 year
  To evaluate the change of quantity of circulating tumor DNA during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Mosser, PUPH, Principal Investigator — Rennes University Hospital
Locations (1):
- CHU, Rennes, France